CLINICAL TRIAL: NCT02911506
Title: Sleep Quality in Intensive Care Unit Patients at High Risk of Extubation Failure
Acronym: WEAN SLEEP 2
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WEAN SLEEP 2
Record Dates: First submitted 2016-09-14; First posted 2016-09-22 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Sleep Quality; Extubation Failure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: Polysomnography

SUMMARY:
The aim of the study is to evaluate the impact of sleep quality on extubation failure rate in intensive care unit patients at high risk.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care units patients intubated for at least 24 hours with at least on of the four following risk factor : aged of 65 years or more, any underlying chronic cardiac or lung disease, mechanical ventilation for more than 7 days.
* aged of 18 years or more

Exclusion Criteria:

* peripheral or central nervous system pathology
* known psychiatric pathology or agitation
* patient with decision of no reintubation
* patient refusal
* clinical worsening before polysomnography ( shock with vasopressors drugs, coma, PaO2/FiO2 ratio < 150 with respiratory distress signs, coma with Glasgow scale <8)
* pregnant or breastfeeding women
* patient under legal guardianship or protection
* patient with no health insurance coverage
* aged < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients, intubated at least 24 hours, at risk of extubation failure
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of sleep quality by polysomnography recording on the extubation day. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France